CLINICAL TRIAL: NCT03487588
Title: An Open-Label Study Assessing Subject Satisfaction With A-101 Hydrogen Peroxide Topical Solution, 40% (w/w) Treatment for Seborrheic Keratoses of the Face, Neck, and Decolletage
Brief Title: An A Study Assessing Subject Satisfaction With A-101 Topical Solution for Seborrheic Keratoses
Acronym: SK-FAN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aclaris Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A-101-SEBK-402
Record Dates: First submitted 2018-03-02; First posted 2018-04-04 (Actual); Results first posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2018-03

CONDITIONS: Seborrheic Keratosis
MeSH Terms: conditions — Keratosis, Seborrheic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- A-101 Topical Solution (Experimental): Open Label Arm
  Interventions: Drug: A-101 Topical Solution

INTERVENTIONS:
Drug: A-101 Topical Solution — A-101 Topical Solution applied Day 1, Day 15 and Day 29

SUMMARY:
This study is an open-label study designed to evaluate subject's satisfaction after treatment of seborrheic keratoses with A-101 40%.

ELIGIBILITY:
Inclusion Criteria:

1. Subject can comprehend and is willing to sign an informed consent for participation in this study.
2. Male or female between the ages of 30 and 75 years old.
3. Subject has 3 eligible Seborrheic Keratoses; 2 target SKs must be on the face, and the additional 1 target SK must be on the neck or decolletage.
4. Subjects must have had cryosurgery for SK removal within the last 6 months and prior to first treatment with A-101 Topical Solution.
5. Target and non-target SKs must not have been previously treated.
6. Subject is in good general health and free of any known disease state or physical condition which, in the investigator's opinion, might impair the evaluation of any target or non-target SK or which exposes the subject to an unacceptable risk by study participation

Exclusion Criteria:

1. Subject has clinically atypical and /or rapidly growing Seborrheic Keratoses.
2. Subject has current systemic malignancy.
3. Subject would require the use of any topical treatment (e.g., moisturizers, sunscreens) to any of the target or non-target SKs 12 hours prior to any study visit.
4. Subject has any current skin disease (e.g., psoriasis, atopic dermatitis, eczema, sun damage), or condition (e.g., sunburn, excessive hair, open wounds) that, in the opinion of the investigator, might put the subject at undue risk by study participation or interfere with the study conduct or evaluations

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2018-11-14 (Actual); Study Completion 2018-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Gordon, MD, Study Director — Aclaris Therapeutics
Locations (3):
- United States (3):
  - Aclaris Investigational Site, Fort Washington, Pennsylvania
  - Aclaris Investigational Site, Knoxville, Tennessee
  - Aclaris Investigational Site, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | A-101 Topical Solution
Started | 41
Completed | 41
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | A-101 Topical Solution
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (6.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 41
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Subject Satisfaction
Description: Subject Satisfaction Questionnaire after treatment with A-101 Topical Solution
Time Frame: Day 113
Measure: Count of Participants; unit: Participants
Arm/Group | A-101 Topical Solution
Number analyzed (Participants) | 41
Participants
  very satisfied (5) | 21
  satsified (4) | 14
  moderately satisfied (3) | 4
  slightly satisfied (2) | 0
  not satisfied at all (1) | 2

2. Secondary Outcome: Effectiveness of Treatment
Description: Effectiveness of treatment as measured by the Physician Lesion Assessment scale. The Physician Lesion Assessment Scale (PLA) is a 4 point scale used by the investigator to assess each subjects SK lesion. PLA=0 (Clear);PLA=1 (Near Clear; not elevated); PLA=2 (Thin;thickness </= 1 mm); PLA=3 (Thick; thickness > 1 mm).
Time Frame: Day 113
Measure: Mean (Standard Deviation); unit: score on a scale (PLA)
Arm/Group | A-101 Topical Solution
Number analyzed (Participants) | 41
score on a scale (PLA) | -2.0 (0.62)

3. Secondary Outcome: Comparison of Physician Lesion Assessment Score (PLA) to Subject Satisfaction
Description: Effectiveness of treatment assessed by PLA (4-point scale) compared to subject reported satisfaction with treatment. The PLA scale is a 4 point scale used by the investigator to assess each subject's SK lesion.
Time Frame: Day 113
Measure: Number; unit: point bi-serial correlation coefficient
Arm/Group | A-101 Topical Solution
Number analyzed (Participants) | 41
point bi-serial correlation coefficient | .318

ADVERSE EVENTS:
Time Frame: 17 weeks; The reporting period for SAEs began when the subject signed the informed consent form. Non serious clinical AEs were collected following the application of the study drug at Visit 2 and continued through Visit 11. All safety reporting (AEs and SAEs) was concluded at Visit 11 (Day 113).
Description: An adverse event (AE) was any untoward medical occurrence in a patient or clinical investigation subject administered a study medication(s) and that did not necessarily have a causal relationship with the study medication.
  Safety summaries by study medication group will include listings by study medication of adverse events incidences within each MedDRA System Organ Class, and changes from pre-application values in vital signs.
Arm/Group | A-101 Topical Solution
All-Cause Mortality (participants affected / at risk) | 0/41
Serious Adverse Events (participants affected / at risk) | 0/41
Other Adverse Events (participants affected / at risk) | 8/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A-101 Topical Solution (N=41)
Eyelid Oedema (Eye disorders) | 2 (2)
Administration site discomfort (General disorders) | 1 (1)
Administration site irritation (General disorders) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Blood cholesterol increased (Investigations) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-06-18): https://cdn.clinicaltrials.gov/large-docs/88/NCT03487588/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-13): https://cdn.clinicaltrials.gov/large-docs/88/NCT03487588/SAP_001.pdf